CLINICAL TRIAL: NCT03962452
Title: Mitochondrial Diseases - Long-read Genome and Transcriptome Sequencing in Cases Unresolved After Short-read Genomics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MiDiSeq
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Rare Diseases; Genetic Predisposition
Keywords: Rare Diseases; Genetic Predisposition; Epigenetic variation; Omics; Genetic variation; Mitochondrial disease; Next Generation Sequencing (NGS)
MeSH Terms: conditions — Rare Diseases; Genetic Predisposition to Disease; Mitochondrial Diseases | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mitochondrial disease (Other): Unresolved index patients with suspected mitochondrial disease
  Interventions: Genetic: Next Generation Sequencing (NGS)

INTERVENTIONS:
Genetic: Next Generation Sequencing (NGS) — Determining the nucleic acid sequence

SUMMARY:
The MiDiSeq project will enroll 20 unresolved index patients with suspected mitochondrial disease prioritized for genomic analysis.

DETAILED DESCRIPTION:
In the MiDiSeq (monocentric, prospective, open-label diagnostic) project, patients with suspected mitochondrial disease prioritized for i) high a priori probability for a genetic basis (e.g. positive family history) as well as availability of (ii) fibroblast cell lines with a biochemically defined phenotype, (iii) parental samples, (iv) short read whole genome and transcriptome datasets and (v) optional additional metabolomics and proteomics data.

The following questions will be leading the project:

i) to systematically benchmark different sequencing technologies to detect genetic and epigenetic variation and their impact on gene regulation.

(ii) to further develop algorithms for integrative analyses of different 'omics datasets.

(iii) to expand the analysis from coding Single-Nucleotide Variants (SNVs) and regulatory mutations to structural variants (SVs), repeat expansions and contractions, low complexity regions and epigenetic signatures.

(iv) to identify novel alterations and disease mechanisms. (v) to gain fundamental new insights into disease mechanisms and cellular biology.

(vi) to improve genetic diagnostics of future rare disease patients and to evaluate personalized therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

Unclear diagnosis Suspected genetic cause of the disease

Exclusion Criteria:

Missing informed consent of the patient/ legal guardian

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
(Epi)Genetic variation | 1 Day
  Number of (Epi)Genetic variation

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Haack, Dr., Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No